CLINICAL TRIAL: NCT05564364
Title: The Effect of Two Different Bikes Exercises on Healthy Knee Joint Cartilage and Lower
Brief Title: The Effect of Bike Exercise on Joint and Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Orhan Güvener, Assistant of Professor, Mersin University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEUTF-FTR-GUVENER-002
Record Dates: First submitted 2022-09-22; First posted 2022-10-03 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Joint; Exercise; Ultrasound; Bicycle
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Controls 1 (Experimental): Healthy individuals participating in the study will be divided into two groups.
  Interventions: Device: Recumbent Bike
- Healthy Controls 2 (Experimental): Healthy individuals participating in the study will be divided into two groups.
  Interventions: Device: Upright Bike

INTERVENTIONS:
Device: Recumbent Bike — The first group will exercise with a recumbent bike for 20 minutes, 3 sessions/week for 6 weeks.
  Arms: Healthy Controls 1
Device: Upright Bike — The first group will exercise with a upright bike for 20 minutes, 3 sessions/week for 6 weeks.
  Arms: Healthy Controls 2

SUMMARY:
The design of our study is a prospective. It is planned to be completed in twenty-four weeks with 34 participants. The main purpose of this study is to examine and compare the effects of two different bike exercises on knee joint and lower extremity muscles by ultrasonographic method.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-35
* Not exercising regularly
* BMI between 18.9-24.9 kg/m2
* Volunteering to participate in the study
* Absence of chronic rheumatic, cardiovascular, neurological, pulmonary or other system diseases that may prevent participation in the exercise program.
* Those who do not have a history of pregnancy, malignant hematological and oncological diseases
* Not smoking
* No musculoskeletal problems of the lower extremity in the last 6 months
* No previous history of lower extremity surgery in the last 1 year

Exclusion Criteria:

* Being outside the age range of 18-35
* Exercising regularly
* Being outside of the BMI 18.9-24.9 kg/m2 range
* Having chronic rheumatic, cardiovascular, neurological, pulmonary or other system diseases that may prevent participation in the exercise program
* Those with a history of pregnancy, malignant hematological and oncological diseases
* Individuals who smoke
* Any musculoskeletal problem of the lower extremity in the last 6 months
* Having a history of lower extremity surgery in the last 1 year

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Baseline knee joint cartilage thickness and muscles thicknesses | Just before first exercises session
  Ultrasonographic measurements will be made using linear probes (5-13 megahertz Logiq P5; GE Medical Systems) .Joint cartillage thickness and lower extremity muscles will measured by ultrasound at baseline.
Knee cartilage thickness and muscles thicknesses after 6 weeks training program | After 6 weeks training program
  Ultrasonographic measurements will be made using linear probes (5-13 megahertz Logiq P5; GE Medical Systems) .Joint cartillage and lower extremity muscles will measured by ultrasound after 6 weeks training program. Joint cartillage thickness and lower extremity muscles will measured by ultrasound after 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Orhan Güvener, MD, Principal Investigator — Mersin University Medical School; Figen Dağ, PhD, Study Chair — Mersin University Medical School
Locations (1):
- Mersin University Department of Physical Medicine and Rehabilitation, Mersin, Turkey (Türkiye)